CLINICAL TRIAL: NCT04478916
Title: Impact of the Comprehensive Geriatric Assessment on the Quality of Life of Elderly Onco-hematologic Patients' Candidates for Complex Antitumoral Therapies: Clinical and Biological Correlatives
Brief Title: Impact of the Comprehensive Geriatric Assessment on the Quality of Life OF Elderly Patients
Acronym: ONCO-AGING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lorenza Scotti (Other)
Responsible Party: Sponsor-Investigator, Lorenza Scotti, Statistician, University of Eastern Piedmont
Organization: University of Eastern Piedmont (Other)
Other Study IDs: ONCO-AGING
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Hematologic Malignancies; Solid Tumor; Elderly Patients
Keywords: Onco-hematologic diseases; Comprehensive Geriatric Assessment (CGA); Screening tool G8; Geriatric Medicine; Precision Medicine; Senescence
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study is designed to evaluate the senescent cells and MDSC; in the peripheral blood of the patients enrolled in the project in 2 time-points: first on basal line (t = 0) and after 12 months or in disease progression. Blood samples (10 ml whole blood) will be collected in Vacutainer EDTA tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Geriatric evaluation Group: Geriatric evaluation of the proportion of elderly patients in which the treatment is modified based on the complete geriatric assessment (CGA)
- Control Group

SUMMARY:
Impact of the Comprehensive Geriatric Assessment on the Quality of Life of elderly onco-hematologic patients' candidates for complex antitumoral therapies: clinical and biological correlatives

DETAILED DESCRIPTION:
The screenings for the next 2 decades indicate an exponential increase in the incidence of neoplastic diseases in the elderly population. In order to successfully balance effectiveness and low toxicity of immunochemotherapy, a treatment personalisation based on an objective evaluation of fitness is therefore needed. The use of geriatric screening is a first step to rationalize decisions in this regard, the G8 tool has demonstrated the ability to identify patients and mostly to objectively separate elderly fragile patients from those who are fit. In that consideration, the individualization of the anticancer treatment based on a Comprehensive Geriatric Assessment (CGA) is desirable in elderly fragile patients with solid or haematological malignancy. Cancer mortality is constantly increasing after 65 years and the consequent increase in life expectancy favour the processes of cellular senescence. In this context G8 fragility assessment will take place in the screening test and by using the EORTC QLQ-C30C questionnaire to assess quality of life (QoL). The evaluation of senescent cells will be done by real-time PCR. Our aims are i) to evaluate the impact of the CGA on the QoL of elderly onco-haematological patients, candidates for complex therapies, that resulted as fragile at the G8 geriatric screening and ii) to evaluate the senescent cells in the peripheral blood of the patients enrolled in the study. The study is expected to contribute to precision medicine management of elderly patients and refine the therapeutic stratifications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 65 years
* Diagnosis of solid or hematologic cancer
* Patients who are candidates for a first line therapy for advanced disease to be treated with biological target drugs, or candidates for integrated radiotherapy
* Patient with G8 scores ≤ 14/17

Exclusion Criteria:

* Patients aged less than 65 years
* Patients who have received or currently in treatment for solid or hematologic cancer
* Patient with G8 scores more than 14/17

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In the present study, only patients aged ≥ 65 years, with diagnosis of solid or hematologic cancer are eligible. Main inclusion criteria are two; i) patients who are candidates for a first line therapy for advanced disease to be treated with biological target drugs, or candidates for integrated radiotherapy; ii) patient with G8 scores ≤ 14/17
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients received planned treatment and CGA evaluated with improvement of good quality of life (QOL) | 12 months after randomization (G8; at screening and every 6 months, QOL; at baseline and every 3 months, CGA; at baseline and every 6 months)
  To assess the impact of the inclusion of the CGA on the quality of life (QOL) of the elderly onco-hematology patient that result frail in the geriatric screening (G8), compared to the clinical practice that does not include the CGA

SECONDARY OUTCOMES:
Number of patients received radiotherapy planned and CGA evaluated with improvement of good quality of life (QOL) | 12 months after randomization (G8; at screening and every 6 months, QOL; at baseline and every 3 months, CGA; at baseline and every 6 months)
  Part of patients receiving radiotherapy will be randomised to be evaluated using CGA compared to control group, the CGA assessment will be done using the status of ADL, IADL, QOL, MNA, SVI, GDS, CIRS, TC, MMSE, CDT, MOCA, RFI, VMD, at baseline and would be re-evaluated after every 6 month and If necessary, an onco-geriatric follow-up will be carried out, for the re-evaluation and further correction of the areas of fragility. A description of the changes of the above scales would also be recorded for the patients
Progression free survival (PFS) | From randomisation (December 2019-December 2022)
  Progression Free Survival (PFS): From the date of diagnosis to the last follow-up, or to one of the following events: disease progression during treatment, or relapse, or death from any cause
Failure Free Survival (FFS) | From randomisation (December 2019-December 2022)
  Failure Free Survival (FFS). From the date of diagnosis to to any treatment failure including disease progression, or discontinuation of treatment for any reason, (eg, disease progression, toxicity, patient preference, initiation of new treatment), or death from any cause
Occurrence of dose reductions | From randomisation through study completion, an average of 1 year
  Data will be collected by reviewing patients medical charts
Overall Survival (OS) | From randomisation (December 2019-December 2022)
  From the date of diagnosis to the last patient last visit

OTHER OUTCOMES:
Senescent cells role in interfering with the planned therapy | 2019-From randomisation until 12 months or until disease progression
  Senescent cells levels and their role in interfering with the planned therapy and the outcome of disease prognosis, PFS, OS. and the correlation between senescent cells level with the results of patients QOL, CGA and G8

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Alessandra Gennari, Principal Investigator — Department of Translational Medicine, Università del Piemonte Orientale
Locations (1):
- Università del Piemonte Orientale - Azienda Ospedliero-Universitaria Maggiore della Carita', Novara, Italy

REFERENCES:
- [Derived] Mahmoud AM, Biello F, Maggiora PM, Bruna R, Burrafato G, Cappelli M, Varughese F, Martini V, Platini F, Deambrogi C, Patriarca A, Nicolosi M, Vachanaram AR, Pisani C, Ferrara E, Catania E, Azzolina D, Barone-Adesi F, Krengli M, Gaidano G, Gennari A. A randomized clinical study on the impact of Comprehensive Geriatric Assessment (CGA) based interventions on the quality of life of elderly, frail, onco-hematologic patients candidate to anticancer therapy: protocol of the ONCO-Aging study. BMC Geriatr. 2021 May 19;21(1):320. doi: 10.1186/s12877-021-02237-3. PMID 34011271